CLINICAL TRIAL: NCT04551430
Title: A Randomized Phase II Trial of Cabozantinib Combined With PD-1 and CTLA-4 Inhibition in Metastatic Soft Tissue Sarcoma
Brief Title: Cabozantinib Combined With PD-1 and CTLA-4 Inhibition in Metastatic Soft Tissue Sarcoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Exelixis (Industry); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 202011041
Record Dates: First submitted 2020-09-01; First posted 2020-09-16 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Metastatic Soft-tissue Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — cabozantinib; Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cohort A: Cabozantinib (Experimental): Patients randomized to Cohort A will take cabozantinib at a dose of 60 mg by mouth once each day of each 28-day cycle. Treatment may continue indefinitely. At time of progression, patients will continue on cabozantinib daily but will reduce their dose to 40 mg. They will cross over into Cohort B and initiate treatment.
  Interventions: Drug: Cabozantinib
- Cohort B: Cabozantinib + Nivolumab + Ipilimumab (Experimental): -Patients randomized to Cohort B will take cabozantinib at a dose of 40 mg by mouth once each day. Nivolumab will given IV at a dose of 3 mg/kg over approximately 30 minutes every 3 weeks for 4 doses, followed by 480 mg over approximately 30 minutes every 4 weeks until treatment discontinuation. Ipilimumab will be given IV at a dose of 1 mg/kg over approximately 30 minutes every 3 weeks for 4 doses. Treatment may continue for up to 2 years.
  Interventions: Drug: Cabozantinib; Drug: Nivolumab; Drug: Ipilimumab
- Crossover from Cohort A to Cohort B: Cabozantinib + Nivolumab + Ipilimumab (Experimental): -Participants who cross-over from Cohort A into Cohort B will initiate treatment with nivolumab at a dose of 3 mg/kg IV over approximately 30 minutes and ipilimumab at a dose of 1 mg/kg IV over approximately 30 minutes. Nivolumab and ipilimumab will be given every 3 weeks for 4 doses. Nivolumab will then be continued at a dose of 480 mg IV over approximately 30 minutes every 4 weeks, with cabozantinib to continue at 40 mg every day. Treatment may continue for up to 2 years.
  Interventions: Drug: Cabozantinib; Drug: Nivolumab; Drug: Ipilimumab

INTERVENTIONS:
Drug: Cabozantinib — Cabozantinib will be supplied by Exelixis.
Drug: Nivolumab — Nivolumab will be provided free of charge (as investigational supply) by Bristol-Myers Squibb.
  Other Names: Opdivo
  Arms: Cohort B: Cabozantinib + Nivolumab + Ipilimumab; Crossover from Cohort A to Cohort B: Cabozantinib + Nivolumab + Ipilimumab
Drug: Ipilimumab — Ipilimumab will be provided free of charge (as investigational supply) by Bristol-Myers Squibb.
  Other Names: Yervoy
  Arms: Cohort B: Cabozantinib + Nivolumab + Ipilimumab; Crossover from Cohort A to Cohort B: Cabozantinib + Nivolumab + Ipilimumab

SUMMARY:
The hypothesis of this study is that the response rate of soft tissue sarcoma will be improved with the addition of PD-1 and CTLA-4 inhibition to cabozantinib, and that cabozantinib priming will increase the response to nivolumab and ipilimumab.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed soft tissue sarcoma that is metastatic or unresectable.
* Measurable disease defined as lesions that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥ 10 mm with CT scan, as ≥ 20 mm by chest x-ray, or ≥ 10 mm with calipers by clinical exam.
* Refractory to at least one and no more than two lines of therapy, with progression on last line of therapy. Neoadjuvant or adjuvant therapy completed more than one year prior does not count towards these two lines of therapy. Individuals with alveolar soft part sarcoma may enroll without being refractory to at least one line of chemotherapy. Any inappropriate therapies (ie hormonal therapies) should be discussed with the PI to determine if they are to be counted toward the two lines of therapy.
* At least 18 years of age.
* ECOG performance status ≤ 1
* Normal bone marrow and organ function as defined below:

  * Absolute neutrophil count ≥ 1,500/mm3 without granulocyte colony-stimulating factor support
  * White blood cell count ≥ 2,000/mm3
  * Platelets ≥ 100,000/mm3 without transfusion
  * Hemoglobin ≥ 9.0 g/dL
  * Total bilirubin ≤ 1.5 x IULN (for subjects with Gilbert's disease, ≤ 3.0 x IULN)
  * AST(SGOT), ALT(SGPT), and alkaline phosphatase (ALP) ≤ 3.0 x IULN; ALP ≤ 5.0 x IULN with documented bone metastases
  * Serum albumin ≥ 2.8 g/dl.
  * Serum creatinine ≤ 1.5x IULN or calculated creatinine clearance ≥ 40 mL/min by MDRD
  * Urine protein/creatinine ration (UPCR) ≤ 1 mg/mg (≤ 113.2 mg/mmol)
  * PT/INR or PTT < 1.3 x IULN (within 7 days before first dose of study treatment, if not receiving any anticoagulation therapy)
* Corrected QT interval calculated by the Fridericia formula (QTcF) ≤ 500 ms (by ECG within 14 days before the first dose of study treatment).
* Lesion amenable to biopsy for assessment of PD-L1 expression if no archival tissue is available
* Recover to baseline or ≤ grade 1 from toxicities related to any prior treatments, unless AE(s) are clinically non-significant and/or stable on supportive therapy.
* The effects of cabozantinib on the developing human fetus are unknown. For this reason, women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry, for the duration of study participation, and for 5 months after the last dose of study treatment. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of the study, and for at least 7 months after the last dose of study treatment.
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria:

* Translocation-driven sarcoma except for ASPS
* Previous treatment with cabozantinib or a PD-1 inhibitor (eg, cemiplimab, nivolumab, pembrolizumab), PD-L1 inhibitor (eg, atezolizumab, avelumab, durvalumab), or CTLA-4 inhibitor (eg, ipilimumab).
* A history of other malignancy with the exception of malignancies for which all treatment was completed at least 2 years before registration and the patient has no evidence of disease. Exceptions include basal cell or squamous cell carcinoma of the skin which were treated with local resection only or carcinoma in situ of the cervix, or other tumors discussed with the study PI.
* Currently receiving any other investigational agents.
* Known brain metastases. Patients with known brain metastases must be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* Receipt of any type of small molecule kinase inhibitor (including investigational kinase inhibitor) within 2 weeks before first dose of study treatment.
* Receipt of any type of cytotoxic, biologic or other systemic anticancer therapy (including investigational) within 4 weeks before first dose of study treatment.
* Concomitant anticoagulation with coumarin agents (e.g., warfarin), direct thrombin inhibitors (e.g., dabigatran), direct factor Xa inhibitor betrixaban, or platelet inhibitors (e.g., clopidogrel). Allowed anticoagulants are the following:

  * Prophylactic use of low-dose aspirin for cardio-protection (per local applicable guidelines) and low dose low molecular weight heparins (LMWH).
  * Therapeutic doses of LMWH or anticoagulation with direct factor Xa inhibitors rivaroxaban, edoxaban, or apixaban in subjects without known brain metastases who are on a stable dose of the anticoagulant for at least 1 week before first dose of study treatment without clinically significant hemorrhagic complications from the anticoagulation regimen or the tumor.
* Radiation therapy for bone metastasis within 2 weeks, any other radiation therapy within 4 weeks before first dose of study treatment. Systemic treatment with radionuclides within 6 weeks before the first dose of study treatment. Subjects with clinically relevant ongoing complications from prior radiation therapy are not eligible.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to cabozantinib, nivolumab, ipilimumab, or other agents used in the study.
* Inability to swallow tablets.
* The subject has uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions:

  * Cardiovascular disorders:

    * Congestive heart failure New York Heart Association Class 3 or 4, unstable angina pectoris, serious cardiac arrhythmias.
    * Uncontrolled hypertension defined as sustained blood pressure (BP) > 140 mm Hg systolic or > 90 mm Hg diastolic despite optimal antihypertensive treatment.
    * Stroke (including transient ischemic attack [TIA]), myocardial infarction (MI), or other ischemic event, or thromboembolic event (e.g., deep venous thrombosis, pulmonary embolism) within 6 months before first dose of study treatment.

      * Subjects with a diagnosis of incidental, subsegmental PE or DVT within 6 months are allowed if stable, asymptomatic, and treated with anticoagulation for at least 1 week before first dose of study treatment.
  * Gastrointestinal (GI) disorders including those associated with a high risk of perforation or fistula formation:

    * The subject has evidence of tumor invading the GI tract, active peptic ulcer disease, inflammatory bowel disease (e.g., Crohn's disease), diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis, acute pancreatitis, acute obstruction of the pancreatic duct or common bile duct, or gastric outlet obstruction.
    * Abdominal fistula, GI perforation, bowel obstruction, or intra-abdominal abscess within 6 months before first dose.
    * Note: Complete healing of an intra-abdominal abscess must be confirmed before first dose.
  * Clinically significant hematuria, hematemesis, or hemoptysis of > 0.5 teaspoon (2.5 ml) of red blood, or other history of significant bleeding (eg, pulmonary hemorrhage) within 12 weeks before first dose.
  * Cavitating pulmonary lesion(s) or known endotracheal or endobronchial disease manifestation.
  * Lesions invading or encasing any major blood vessels.
  * Other clinically significant disorders that would preclude safe study participation.

    * Serious non-healing wound/ulcer/bone fracture.
    * Uncompensated/symptomatic hypothyroidism.
    * Moderate to severe hepatic impairment (Child-Pugh B or C)
* Any active, known, or suspected autoimmune disease Note: subjects with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
* Any condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of randomization Note: inhaled, intranasal, intra-articular, or topical steroids are permitted. Adrenal replacement steroid doses > 10 mg daily prednisone equivalent are permitted in the absence of active autoimmune disease. Transient short-term use of systemic corticosteroids for allergic conditions (e.g. contrast allergy) is also allowed.
* Active infection requiring systemic treatment. Acute or chronic hepatitis B or C infection, known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness, or known positive test for tuberculosis infection
* History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, or evidence of active pneumonitis on screening chest CT scan
* Malabsorption syndrome
* Requirement for hemodialysis or peritoneal dialysis
* History of solid organ or allogeneic stem cell transplant.
* Major surgery (e.g. laparoscopic nephrectomy, GI surgery removal or biopsy of brain metastasis) within 2 weeks before first dose of study treatment. Minor surgeries within 10 days before first dose of study treatment. Subjects must have complete wound healing from major surgery or minor surgery before first dose of study treatment. Patients with clinically relevant ongoing complications from prior surgery are not eligible.
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative pregnancy test within 15 days of study entry. Women of childbearing potential are defined as premenopausal females capable of becoming pregnant (i.e., females who have had any evidence of menses in the past 12 months, with the exception of those who had prior hysterectomy). However, women who have been amenorrheic for 12 or more months are still considered to be of childbearing potential if the amenorrhea is possibly due to prior chemotherapy, antiestrogens, low body weight, ovarian suppression, or other reasons
* Administration of a live, attenuated vaccine within 30 days prior to randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2021-01-05 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2029-02-01 (Estimated)

PRIMARY OUTCOMES:
Radiographic response rate by RECIST 1.1 | From start of treatment until disease progression/recurrence or the date of subsequent therapy (estimated to be 24 months)
  * Response rate = proportion of participants who achieve complete response or partial response
  * Complete response: Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Disappearance of all non-target lesions and normalization of tumor marker level. All lymph nodes must be non-pathological in size (<10 mm short axis).
  * Partial response: At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.

SECONDARY OUTCOMES:
Clinical benefit rate | Through end of treatment (estimated to be 24 months)
  -A confirmed clinical benefit is defined to be either a CR or PR noted as the objective status on 2 consecutive evaluations at least 4 weeks apart or a confirmed SD at two consecutive tumor assessments at least 3 months apart. The CBR will be estimated by the number of patients with confirmed clinical benefit divided by the total number of evaluable patients
Progression-free survival | Up to 3 years from end of treatment
  * PFS is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first.
  * Progressive disease: Appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions. Unequivocal progression should not normally trump target lesion status. It must be representative of overall disease status change, not a single lesion increase.
  * Patients will be censored at time of subsequent treatment regardless of response
Overall survival | Up to 5 years from end of treatment
  * Defined as from date of treatment start to date of death or date of last follow up if alive
  * Patients will be censored at time of subsequent treatment regardless of response
Response rate to ipilimumab + nivolumab after cabozantinib priming | Through end of treatment (estimated to be 24 months)
  * Response rate = proportion of participants who achieve complete response or partial response
  * Complete response: Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Disappearance of all non-target lesions and normalization of tumor marker level. All lymph nodes must be non-pathological in size (<10 mm short axis).
  * Partial response: At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Change in quality of life as measured by FACT-G7 | Baseline, day 1 of each cycle (each cycle is 4 weeks), and at time of disease progression (estimated to be up to 5 years)
  * 7 statements with answers ranging from 0=Not at all to 4=Very much. The higher the score, the better the quality of life
  * The sum of the item scores will be multiplied by the number of items in the subscale then divided by the number of items answered. This will produce the total score.
Radiographic response rate by iRECIST | From start of treatment until disease progression/recurrence or the date of subsequent therapy (estimated to be 24 months)
  Response rate = proportion of participants who achieve immune complete response or immune partial response

CONTACTS AND LOCATIONS:
Overall Officials: Mia Weiss, M.D., Principal Investigator — Washington University School of Medicine
Locations (4):
- United States (4):
  - Stanford University Medical Center, Stanford, California
  - University of Colorado, Aurora, Colorado
  - Washington University School of Medicine, St Louis, Missouri
  - Abramson Cancer Center at Pennsylvania Hospital, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu